CLINICAL TRIAL: NCT05610956
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Empagliflozin in Patients With Ulcerative Colitis
Brief Title: Evaluate the Possible Efficacy and Safety of Empagliflozin in Patient With Ulcerative Colitis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Youmna Hamdy, pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: empagliflozin in UC
Record Dates: First submitted 2022-10-31; First posted 2022-11-09 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: parallel randomized controlled
Who Masked: Participant, Investigator
Masking Description: double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo group (Placebo Comparator): Patients will receive conventional treatment only (corticosteroids +immune suppressive +amino salicylic acid) for 4 months.
  Interventions: Drug: conventional treatment
- empagliflozin group (Experimental): Patients will receive conventional treatment (corticosteroids +immune suppressive + aminosalicylic acid) and empagliflozin (0.4 - 0.5mg/kg/day) orally (maximum dose 25mg per day)for 4months.
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — Patients will receive empagliflozin (0.4 - 0.5mg/kg/day) orally (maximum dose 25mg per day)and conventional treatment (corticosteroids +immune suppressive + aminosalicylic acid)for 4 months.
  Arms: empagliflozin group
Drug: conventional treatment — conventional treatment (corticosteroids +immune suppressive + aminosalicylic acid)for 4 months
  Arms: placebo group

SUMMARY:
•This study will be a randomized, controlled, parallel study. .To demonstrate the efficacy of empagliflozin and clinical improvement in patients of mild to moderate UC using the Montreal classification of severity of ulcerative colitis.

DETAILED DESCRIPTION:
* It will be conducted on 60 patients having with mild to moderate degree UC divided into two groups:

  1. Group 1 (n=30): Patients will receive conventional treatment only (corticosteroids +immune suppressive +amino salicylic acid).
  2. Group 2 (n=30): Patients will receive conventional treatment (corticosteroids +immune suppressive + aminosalicylic acid) and empagliflozin (0.4 - 0.5mg/kg/day) orally (maximum dose 25mg per day).
* The patient will be selected from the Gastroenterology and Endoscopy Unit, Internal Medicine.

  . All patients will be subjected to the following:
* Complete history taking.
* Colonoscopy with intubation of the ileum and biopsies of affected and unaffected areas should be obtained to confirm the diagnosis of UC.
* Blood sample collection to assess:

A) Routine Laboratory tests

1. Complete blood picture (CBC).
2. Liver functions (ALT, AST, Total and Direct Bilirubin).
3. Kidney functions tests (Urea, serum creatinine).
4. C-reactive protein.
5. Fasting blood glucose.
6. Urine analysis. B) Specific Laboratory tests

1. Tumor necrosis factor alpha (TNF-α). 2. Adenosine monophosphate activate protein kinase (AMPK). 3. Fecal calprotectin. All patients will be assessed at baseline and after 4 months of therapy for all parameters

ELIGIBILITY:
Inclusion Criteria:

•Patients with mild to moderate UC are diagnosed by history, clinical signs according to the Montreal classification of severity of ulcerative colitis and( Endoscopy, and biopsy) to establish the chronicity of inflammation and to exclude other causes of colitis.

Exclusion Criteria:

* Other inflammatory bowel diseases (CD).
* History of serious hypersensitivity to empagliflozin or any component of the formulation.
* Patients on dialysis.
* Severe renal impairment (eGFR <20 ml/minute/1.73m2) .
* Chronic urinary tract infection.
* Chronic genital infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
clinical improvement of patients of mild to moderate UC using using the Montreal classification of severity of ulcerative colitis. | 4months
  difference between the two groups in (number of stool per day+prescence of fever +present of systemic toxicity+hemoglibin +ESR)

SECONDARY OUTCOMES:
expression of TNFalpha | 4months
  difference between the two groups in TNFalpha
expression of Adenosine monophosphate activated protein kinase (AMPK ). | 4months
  difference between the two groups in Adenosine monophosphate activated protein kinase (AMPK )
expression of Fecal calprotectin | 4months
  difference between the two groups in fecal calprotectin

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology and Endoscopy Unit, Internal Medicine Department, Tanta University Hospital., Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Karle EJ, Gehring F, Trautner K. [Cariogenic properties of various snacks in animal experiments]. Dtsch Zahnarztl Z. 1977 Sep;32(9):741-3. German. PMID 269076
- [Background] Rubin DT, Huo D, Kinnucan JA, Sedrak MS, McCullom NE, Bunnag AP, Raun-Royer EP, Cohen RD, Hanauer SB, Hart J, Turner JR. Inflammation is an independent risk factor for colonic neoplasia in patients with ulcerative colitis: a case-control study. Clin Gastroenterol Hepatol. 2013 Dec;11(12):1601-8.e1-4. doi: 10.1016/j.cgh.2013.06.023. Epub 2013 Jul 17. PMID 23872237
- [Background] Gasche C, Scholmerich J, Brynskov J, D'Haens G, Hanauer SB, Irvine EJ, Jewell DP, Rachmilewitz D, Sachar DB, Sandborn WJ, Sutherland LR. A simple classification of Crohn's disease: report of the Working Party for the World Congresses of Gastroenterology, Vienna 1998. Inflamm Bowel Dis. 2000 Feb;6(1):8-15. doi: 10.1097/00054725-200002000-00002. PMID 10701144
- [Background] Colman RJ, Rubin DT. Histological inflammation increases the risk of colorectal neoplasia in ulcerative colitis: a systematic review. Intest Res. 2016 Jul;14(3):202-10. doi: 10.5217/ir.2016.14.3.202. Epub 2016 Jun 27. PMID 27433141
- [Background] Esmat S, El Nady M, Elfekki M, Elsherif Y, Naga M. Epidemiological and clinical characteristics of inflammatory bowel diseases in Cairo, Egypt. World J Gastroenterol. 2014 Jan 21;20(3):814-21. doi: 10.3748/wjg.v20.i3.814. PMID 24574754
- [Background] Jess T, Frisch M, Simonsen J. Trends in overall and cause-specific mortality among patients with inflammatory bowel disease from 1982 to 2010. Clin Gastroenterol Hepatol. 2013 Jan;11(1):43-8. doi: 10.1016/j.cgh.2012.09.026. Epub 2012 Sep 27. PMID 23022699
- [Background] Regueiro M, Greer JB, Szigethy E. Etiology and Treatment of Pain and Psychosocial Issues in Patients With Inflammatory Bowel Diseases. Gastroenterology. 2017 Feb;152(2):430-439.e4. doi: 10.1053/j.gastro.2016.10.036. Epub 2016 Nov 2. PMID 27816599
- [Background] MacDermott RP, Sanderson IR, Reinecker HC. The central role of chemokines (chemotactic cytokines) in the immunopathogenesis of ulcerative colitis and Crohn's disease. Inflamm Bowel Dis. 1998 Feb;4(1):54-67. doi: 10.1097/00054725-199802000-00009. PMID 9552229
- [Background] Greenstein AJ, Sachar DB, Gibas A, Schrag D, Heimann T, Janowitz HD, Aufses AH Jr. Outcome of toxic dilatation in ulcerative and Crohn's colitis. J Clin Gastroenterol. 1985 Apr;7(2):137-43. doi: 10.1097/00004836-198504000-00007. PMID 4008909
- [Background] Jalan KN, Sircus W, Card WI, Falconer CW, Bruce CB, Crean GP, McManus JP, Small WP, Smith AN. An experience of ulcerative colitis. I. Toxic dilation in 55 cases. Gastroenterology. 1969 Jul;57(1):68-82. No abstract available. PMID 5305933
- [Background] Bedine MS. Textbook of gastroenterology. Gastroenterology. 2000 May;118(5):984-5. doi: 10.1016/s0016-5085(00)70191-0. No abstract available. PMID 10784603
- [Background] Bernstein CN, Wajda A, Blanchard JF. The incidence of arterial thromboembolic diseases in inflammatory bowel disease: a population-based study. Clin Gastroenterol Hepatol. 2008 Jan;6(1):41-5. doi: 10.1016/j.cgh.2007.09.016. Epub 2007 Dec 11. PMID 18063423
- [Background] Merigo F, Brandolese A, Facchin S, Missaggia S, Bernardi P, Boschi F, D'Inca R, Savarino EV, Sbarbati A, Sturniolo GC. Glucose transporter expression in the human colon. World J Gastroenterol. 2018 Feb 21;24(7):775-793. doi: 10.3748/wjg.v24.i7.775. PMID 29467549
- [Background] Zhou H, Wang S, Zhu P, Hu S, Chen Y, Ren J. Empagliflozin rescues diabetic myocardial microvascular injury via AMPK-mediated inhibition of mitochondrial fission. Redox Biol. 2018 May;15:335-346. doi: 10.1016/j.redox.2017.12.019. Epub 2017 Dec 30. PMID 29306791
- [Background] Iannantuoni F, M de Maranon A, Diaz-Morales N, Falcon R, Banuls C, Abad-Jimenez Z, Victor VM, Hernandez-Mijares A, Rovira-Llopis S. The SGLT2 Inhibitor Empagliflozin Ameliorates the Inflammatory Profile in Type 2 Diabetic Patients and Promotes an Antioxidant Response in Leukocytes. J Clin Med. 2019 Nov 1;8(11):1814. doi: 10.3390/jcm8111814. PMID 31683785